CLINICAL TRIAL: NCT00287781
Title: A Double Blind Randomized Controlled of Placebo and Nebulized Lidocaine for Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kern Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: #04028
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Migraine Headache
Keywords: Migraine; Lidocaine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
Migraine headaches have previously been shown to be responsive to intranasal lidocaine in a small study. Using a nebulizer to administer the drug would improve the feasibility of using the treatment. It would also spare the patient narcotics with their attendant side effects. Because of the potential for placebo effect a placebo control is necessary in this study.

ELIGIBILITY:
Inclusion Criteria:

* Meets IHS criteria for migraine

Exclusion Criteria:

* Pregnant
* Breast feeding
* Allergic to Lidocaine
* Worst or first Headache
* Abnormal neurological exam
* Substance abuse within 6 months
* Cardiac, liver or pulmonary disease
* Participation n another study within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2002-01; Study Completion 2006-04

PRIMARY OUTCOMES:
Resolution of symptoms

SECONDARY OUTCOMES:
Improvement in 10 point pain score

CONTACTS AND LOCATIONS:
Overall Officials: Rick McPheeters, DO FAAEM, Principal Investigator — Kern Medical Center UCLA
Locations (1):
- Kern Medical Center, Bakersfield, California, United States